CLINICAL TRIAL: NCT03094975
Title: A Multicenter Registry Study of Aneurysmal Subarachnoid Hemorrhage
Brief Title: A Multicenter Registry Study of Aneurysmal SAH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jian-min Liu (Other)
Responsible Party: Sponsor-Investigator, Jian-min Liu, Director, Changhai Hospital
Organization: Changhai Hospital (Other)
Other Study IDs: CHEC2017-022
Record Dates: First submitted 2017-03-11; First posted 2017-03-29 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Time Delay
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Firstly, this study aims at clarifying the current situation of Emergency treatment of aneurysmal subarachnoid hemorrhage (SAH) in China, and analyzing the influencing factors contributing to transport delay, so as to improve the efficiency of emergency treatment; Secondly, comparison and analysis of different surgical treatment of aneurysmal SAH would be undertook, so as to improve the diagnosis and treatment of aneurysmal SAH.

ELIGIBILITY:
Inclusion Criteria:

* patients presented with subarachnoid hemorrhage on CT or lumbar puncture.
* the intracranial hemorrhage was caused by rupture of aneurysm and was confirmed on CTA、MRA or DSA.
* patients willing to participate in this clinical trial and attach to regular follow up.

Exclusion Criteria:

* intracranial aneurysm correlating to AVM.
* dissection, false, traumatic and infectious aneurysms.
* the rupture of the aneurysm can not be confirmed on CTA、MRA or DSA.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients presented with subarachnoid hemorrhage and diagnosed with ruptured aneurysm at all age.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Door to Puncture | the time interval would be noted and be analyzed through study completion, an average of 6 months.
  the time interval between admission to hospital and puncture

SECONDARY OUTCOMES:
Door to CT | the time interval would be noted and be analyzed through study completion, an average of 6 months.
  the time interval between admission to hospital and time of CT performed

OTHER OUTCOMES:
Onset to Door | the time interval would be noted and be analyzed through study completion, an average of 6 months.
  the time interval between onset of symptom and admission to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, MD., Principal Investigator — Changhai Hospital
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Rooij NK, Linn FH, van der Plas JA, Algra A, Rinkel GJ. Incidence of subarachnoid haemorrhage: a systematic review with emphasis on region, age, gender and time trends. J Neurol Neurosurg Psychiatry. 2007 Dec;78(12):1365-72. doi: 10.1136/jnnp.2007.117655. Epub 2007 Apr 30. PMID 17470467
- [Result] Kozak N, Hayashi M. Trends in the incidence of subarachnoid hemorrhage in Akita Prefecture, Japan. J Neurosurg. 2007 Feb;106(2):234-8. doi: 10.3171/jns.2007.106.2.234. PMID 17410705
- [Result] Molyneux A, Kerr R, Stratton I, Sandercock P, Clarke M, Shrimpton J, Holman R; International Subarachnoid Aneurysm Trial (ISAT) Collaborative Group. International Subarachnoid Aneurysm Trial (ISAT) of neurosurgical clipping versus endovascular coiling in 2143 patients with ruptured intracranial aneurysms: a randomised trial. Lancet. 2002 Oct 26;360(9342):1267-74. doi: 10.1016/s0140-6736(02)11314-6. PMID 12414200
- [Result] Johnston SC, Selvin S, Gress DR. The burden, trends, and demographics of mortality from subarachnoid hemorrhage. Neurology. 1998 May;50(5):1413-8. doi: 10.1212/wnl.50.5.1413. PMID 9595997
- [Result] Bian LH, Liu YF, Nichols LT, Wang CX, Wang YL, Liu GF, Wang WJ, Zhao XQ. Epidemiology of subarachnoid hemorrhage, patterns of management, and outcomes in China: a hospital-based multicenter prospective study. CNS Neurosci Ther. 2012 Nov;18(11):895-902. doi: 10.1111/cns.12001. Epub 2012 Sep 12. PMID 22966850
- [Result] Cross DT 3rd, Tirschwell DL, Clark MA, Tuden D, Derdeyn CP, Moran CJ, Dacey RG Jr. Mortality rates after subarachnoid hemorrhage: variations according to hospital case volume in 18 states. J Neurosurg. 2003 Nov;99(5):810-7. doi: 10.3171/jns.2003.99.5.0810. PMID 14609158
- [Result] Shea AM, Reed SD, Curtis LH, Alexander MJ, Villani JJ, Schulman KA. Characteristics of nontraumatic subarachnoid hemorrhage in the United States in 2003. Neurosurgery. 2007 Dec;61(6):1131-7; discussion 1137-8. doi: 10.1227/01.neu.0000306090.30517.ae. PMID 18162891
- [Result] Li H, Pan R, Wang H, Rong X, Yin Z, Milgrom DP, Shi X, Tang Y, Peng Y. Clipping versus coiling for ruptured intracranial aneurysms: a systematic review and meta-analysis. Stroke. 2013 Jan;44(1):29-37. doi: 10.1161/STROKEAHA.112.663559. Epub 2012 Dec 13. PMID 23238862
- [Result] Darsaut TE, Raymond J. Barrow Ruptured Aneurysm Trial: 3-year results. J Neurosurg. 2013 Dec;119(6):1642-4. doi: 10.3171/2013.5.JNS13917. Epub 2013 Aug 30. No abstract available. PMID 23991842
- [Result] Dacks PA, Armstrong JJ, Brannan SK, Carman AJ, Green AM, Kirkman MS, Krakoff LR, Kuller LH, Launer LJ, Lovestone S, Merikle E, Neumann PJ, Rockwood K, Shineman DW, Stefanacci RG, Velentgas P, Viswanathan A, Whitmer RA, Williamson JD, Fillit HM. A call for comparative effectiveness research to learn whether routine clinical care decisions can protect from dementia and cognitive decline. Alzheimers Res Ther. 2016 Aug 20;8:33. doi: 10.1186/s13195-016-0200-3. PMID 27543171